CLINICAL TRIAL: NCT03733912
Title: To Investigate the Effect of Plasticizers on the Pregnancy in Vitro Fertilization Cycles
Brief Title: Plasticizers and in Vitro Fertilization Outcomes
Status: Completed | Type: Observational
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Dr., Kaohsiung Veterans General Hospital.
Other Study IDs: VGHKS18-CT3-09
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Fertilization in Vitro
MeSH Terms: interventions — Diethylhexyl Phthalate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnancy: Infertile women undergoing in vitro fertilization cycle got pregnancy successfully. The pregnancy persisted over 12 weeks.
  Interventions: Other: Phthalate metabolites measurement
- Non-pregnancy: Infertile women undergoing in vitro fertilization cycle failed to reach pregnancy.
  Interventions: Other: Phthalate metabolites measurement

INTERVENTIONS:
Other: Phthalate metabolites measurement — To measure phthalate metabolites of urine and house dust in Pregnancy and Non-pregnancy groups
  Other Names: diethylhexyl phthalate

SUMMARY:
To investigate the effect of Plasticizer metabolites concentration on the in vitro fertilization outcomes

DETAILED DESCRIPTION:
This study was conducted in a medical center in southern Taiwan. 80 infertile female patients, aged 30 to 40 years old with normal ovarian function, receiving IVF treatment in the infertility outpatient were enrolled in this study. The participates were divided into two groups: successful pregnancy in the IVF cycle (n = 40) and non-pregnancy in the IVF cycle (n = 40). After getting the consent of the patients, we plan to do a questionnaire survey. Additionally, environmental dust and urine were sampled and analyzed the concentration of plasticizers metabolites.The aim of this study is to investigate the effect of Plasticizer metabolites concentration on the in vitro fertilization outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women undergoing in vitro fertilization cycles
* Normal ovarian reserve (AMH > 1.0 and AFC ≧ 5)

Exclusion Criteria:

* Daily homestay time > 12 hrs
* Diminished ovarian reserve (AMH ≦ 1.0 or AFC<5)
* Oophorectomy
* Gynecologic cancer patients
* Severe male infertility

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: This study was conducted in a medical center in southern Taiwan. 80 infertile female patients, aged 30 to 40 years old with normal ovarian function, receiving IVF treatment in the infertility outpatient were enrolled in this study. The participates were divided into two groups: successful pregnancy in the IVF cycle (n = 40) and non-pregnancy in the IVF cycle (n = 40). After getting the consent of the patients, we plan to do a questionnaire survey. Additionally, environmental dust and urine were sampled and analyzed the concentration of plasticizers metabolites.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Phthalate of urine | through study completion, an average of 1 year
  Phthalate metabolites concentrations

SECONDARY OUTCOMES:
Phthalate of environmental dust | through study completion, an average of 1 year
  Phthalate metabolites concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, PhD, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messerlian C, Souter I, Gaskins AJ, Williams PL, Ford JB, Chiu YH, Calafat AM, Hauser R; Earth Study Team. Urinary phthalate metabolites and ovarian reserve among women seeking infertility care. Hum Reprod. 2016 Jan;31(1):75-83. doi: 10.1093/humrep/dev292. Epub 2015 Nov 15. PMID 26573529
- [Background] Chen ML, Chen JS, Tang CL, Mao IF. The internal exposure of Taiwanese to phthalate--an evidence of intensive use of plastic materials. Environ Int. 2008 Jan;34(1):79-85. doi: 10.1016/j.envint.2007.07.004. Epub 2007 Aug 31. PMID 17765308
- [Background] Jurewicz J, Hanke W. Exposure to phthalates: reproductive outcome and children health. A review of epidemiological studies. Int J Occup Med Environ Health. 2011 Jun;24(2):115-41. doi: 10.2478/s13382-011-0022-2. Epub 2011 May 19. PMID 21594692
- [Background] Koch HM, Lorber M, Christensen KL, Palmke C, Koslitz S, Bruning T. Identifying sources of phthalate exposure with human biomonitoring: results of a 48h fasting study with urine collection and personal activity patterns. Int J Hyg Environ Health. 2013 Nov;216(6):672-81. doi: 10.1016/j.ijheh.2012.12.002. Epub 2013 Jan 18. PMID 23333758
- [Background] Shea KM; American Academy of Pediatrics Committee on Environmental Health. Pediatric exposure and potential toxicity of phthalate plasticizers. Pediatrics. 2003 Jun;111(6 Pt 1):1467-74. doi: 10.1542/peds.111.6.1467. PMID 12777573
- [Background] Becker K, Seiwert M, Angerer J, Heger W, Koch HM, Nagorka R, Rosskamp E, Schluter C, Seifert B, Ullrich D. DEHP metabolites in urine of children and DEHP in house dust. Int J Hyg Environ Health. 2004 Oct;207(5):409-17. doi: 10.1078/1438-4639-00309. PMID 15575555
- [Background] Du YY, Guo N, Wang YX, Hua X, Deng TR, Teng XM, Yao YC, Li YF. Urinary phthalate metabolites in relation to serum anti-Mullerian hormone and inhibin B levels among women from a fertility center: a retrospective analysis. Reprod Health. 2018 Feb 23;15(1):33. doi: 10.1186/s12978-018-0469-8. PMID 29471860
- [Background] Wu H, Ashcraft L, Whitcomb BW, Rahil T, Tougias E, Sites CK, Pilsner JR. Parental contributions to early embryo development: influences of urinary phthalate and phthalate alternatives among couples undergoing IVF treatment. Hum Reprod. 2017 Jan;32(1):65-75. doi: 10.1093/humrep/dew301. Epub 2016 Dec 7. PMID 27927842
- [Background] Vabre P, Gatimel N, Moreau J, Gayrard V, Picard-Hagen N, Parinaud J, Leandri RD. Environmental pollutants, a possible etiology for premature ovarian insufficiency: a narrative review of animal and human data. Environ Health. 2017 Apr 7;16(1):37. doi: 10.1186/s12940-017-0242-4. PMID 28388912
- [Background] Minguez-Alarcon L, Gaskins AJ. Female exposure to endocrine disrupting chemicals and fecundity: a review. Curr Opin Obstet Gynecol. 2017 Aug;29(4):202-211. doi: 10.1097/GCO.0000000000000373. PMID 28557831
- [Background] Richardson MC, Guo M, Fauser BC, Macklon NS. Environmental and developmental origins of ovarian reserve. Hum Reprod Update. 2014 May-Jun;20(3):353-69. doi: 10.1093/humupd/dmt057. Epub 2013 Nov 27. PMID 24287894
- [Result] Hauser R, Gaskins AJ, Souter I, Smith KW, Dodge LE, Ehrlich S, Meeker JD, Calafat AM, Williams PL; EARTH Study Team. Urinary Phthalate Metabolite Concentrations and Reproductive Outcomes among Women Undergoing in Vitro Fertilization: Results from the EARTH Study. Environ Health Perspect. 2016 Jun;124(6):831-9. doi: 10.1289/ehp.1509760. Epub 2015 Nov 6. PMID 26545148
- [Result] Wu H, Olmsted A, Cantonwine DE, Shahsavari S, Rahil T, Sites C, Pilsner JR. Urinary phthalate and phthalate alternative metabolites and isoprostane among couples undergoing fertility treatment. Environ Res. 2017 Feb;153:1-7. doi: 10.1016/j.envres.2016.11.003. Epub 2016 Nov 19. PMID 27875712